CLINICAL TRIAL: NCT07373431
Title: Biomarkers for Epilepsy Development and the Effect of Physical Exercise in Children With Autism
Acronym: ASD/EP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-03207
Record Dates: First submitted 2026-01-09; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Epilepsy; Autism Spectrum Disorder
Keywords: epilepsy; autism spectrum disorder; Biomarkers; Immunological factors; Circadian rhythm; Cognitive function; Physical activity; Exercise intervention; Seizures
MeSH Terms: conditions — Epilepsy; Autism Spectrum Disorder; Motor Activity; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical activity intervention program (Experimental): Participants will engage in a structured physical exercise program conducted in small groups, 1-3 times per week, over 8-12 weeks. Each session lasts up to 1 hour and includes heart-rate-raising aerobic activities followed by a relaxation period.
  Interventions: Behavioral: Physical activity program

INTERVENTIONS:
Behavioral: Physical activity program — Participants will engage in a structured physical exercise program conducted in small groups, 1-3 times per week, over 8-12 weeks. Each session lasts up to 1 hour and includes heart-rate-raising aerobic activities followed by a relaxation period.

SUMMARY:
This study aims to identify novel biomarkers for epilepsy development in children with autism and to evaluate the effects of physical exercise on these biomarkers and clinical outcomes. Very little is known about epilepsy biomarkers in children with autism, and the risk of developing epilepsy in this population ranges from 5% to 47%. The project focuses on potential signaling pathways, including immunological factors, synaptic proteins, circadian rhythm genes, sleep architecture, and cognitive function.

Children with autism, with or without epilepsy, as well as children with epilepsy, will undergo genetic analyses (exome sequencing) of synaptic and circadian rhythm-related genes, immunological protein profiling, EEG or polysomnography, actigraphy, neuropsychological testing, and physical assessments including coordination, balance, and body awareness. Participants will also engage in a three-month structured physical exercise program. Follow-up assessments will examine the effects of exercise on seizure frequency, biomarker expression, sleep, cognition, and physical abilities.

The study addresses two key research questions: 1) whether biomarkers and physiological measures correlate with seizure occurrence in children with autism, and 2) whether regular physical activity can modulate seizure frequency, biomarker expression, circadian rhythm, sleep, cognitive performance, and physical skills. The findings are expected to improve understanding of the mechanisms underlying epilepsy in autism and inform potential interventions.

DETAILED DESCRIPTION:
The project aims to explore novel biomarkers for the development of epilepsy in children with autism and to evaluate how physical exercise may influence the expression of these biomarkers as well as the severity of epilepsy and autism. Currently, limited knowledge exists within this research field, and the risk of developing epilepsy in individuals with autism varies considerably. One hypothesis is that autism and epilepsy may partly arise from similar genetic alterations in synaptic proteins and exhibit comparable variations in immunological protein levels. Children with autism as well as children with epilepsy also have an increased risk of disrupted circadian rhythm and sleep disturbances, as well as dysfunction in genes regulating circadian rhythms. Physical exercise has been associated with changes in inflammatory responses, epilepsy development, cognitive brain functions, and circadian rhythm/sleep patterns.

The project includes children with autism with or without epilepsy, as well as children with epilepsy, who will:

1. Provide blood samples for genetic analyses (exome sequencing) focusing on synaptic proteins and circadian clock genes. Blood samples will also be collected from both biological parents for comparison. Immunological protein levels will be analyzed in a separate blood sample from the children.
2. Undergo electroencephalography (EEG) or polysomnography (PSG) to assess brain electrical activity during sleep, as well as actigraphy to evaluate circadian rhythm.
3. Undergo neuropsychological testing, including assessments of memory, executive function, and attention, as well as physical tests focusing primarily on coordination, balance, and body awareness.
4. Participate in a physical exercise program for approximately three months.
5. After completion of the physical exercise program, provide follow-up blood samples for immunological protein analyses and undergo repeat EEG or PSG with actigraphy, as well as cognitive and physical testing.

The aim of this study is to explore biomarkers for the development of epilepsy in children with autism and to evaluate the extent to which these signaling pathways, as well as the severity of epilepsy and autism, can be influenced by physical activity. Very little has been published on biomarkers for epilepsy in children with autism. According to previous studies, the risk of developing epilepsy in children with autism ranges from 5% to 47%.

In the present research project, the investigators focus on identifying potential signaling pathways that may serve as biomarkers. These include primarily immunological factors, synaptic proteins, circadian clock genes, sleep architecture, and circadian rhythm. The research group also investigate whether physical exercise can influence the expression of these biomarkers, sleep architecture, cognitive function, physical abilities such as coordination, balance, and body awareness, as well as seizure frequency.

Scientific Research Questions:

1. Can the expression of immunological factors in blood, alterations in synaptic and circadian rhythm genes, circadian rhythm patterns, cognitive function, or EEG changes be correlated with the occurrence of epileptic seizures in children with autism?
2. Can regular physical exercise in children with autism, with or without epilepsy, influence the onset or frequency of epileptic seizures, the expression of immunological factors, circadian rhythm, sleep architecture, cognitive abilities, and physical skills such as balance, coordination, and body awareness?

ELIGIBILITY:
Inclusion Criteria:

* Children aged 10-15 years
* Diagnosed with mild-to-moderate autism spectrum disorder and/or diagnosed with epilepsy

Exclusion Criteria:

* Severe autism spectrum disorder
* Severe cognitive impairment
* Severe ADHD
* Active systemic inflammatory or neurodegenerative disease
* Traumatic brain injury within the past 6 months

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Blood sample collection for genetic and protein analyses | Will be conducted at baseline (time of enrollment) and again 1-3 months after completion of the physical exercise intervention, within 6 months from baseline.
  Participants will provide venous blood samples (maximum 10 mL per occasion, up to 2 occasions) for genetic analyses, focusing on synaptic proteins and circadian clock genes (exome sequencing of approximately 600 genes), as well as protein analyses using ELISA, Western blot, or equivalent techniques to assess immunologically associated proteins, including pro- and anti-inflammatory proteins and cell death-related proteins.
  Biological parents of the children will also provide blood samples for comparison in the genetic analyses. Parental consent for this blood collection will be obtained using a separate consent form.
Actigraphy to evaluate sleep-wake patterns: Sleep latency (minutes) | Will be conducted at baseline (time of enrollment) and again 1-3 months after completion of the physical exercise intervention, within 6 months from baseline.
  Sleep-wake patterns were evaluated using actigraphy. The children were asked to wear an actigraphy watch (MotionWatch 8, CamNtech, UK), which monitors movement and light exposure, for 5-7 days. Sleep latency (minutes) was measured as the duration between the time point the child tries to go to sleep (lights out) and the start of the first block of immobility (presumed fell asleep).
Actigraphy to evaluate sleep-wake patterns: Assumed sleep (hours) | Will be conducted at baseline (time of enrollment) and again 1-3 months after completion of the physical exercise intervention, within 6 months from baseline.
  Actigraphy to evaluate sleep-wake patterns Description: Sleep-wake patterns were evaluated using actigraphy. The children were asked to wear an actigraphy watch (MotionWatch 8, CamNtech, UK), which monitors movement and light exposure, for 5-7 days. Assumed sleep (the sleep period; hours) represents the duration from fell asleep to the end of the last part/block of immobility before getting out of bed (woke up).
Actigraphy to evaluate sleep-wake patterns: Fragmentation Index (index units) | Will be conducted at baseline (time of enrollment) and again 1-3 months after completion of the physical exercise intervention, within 6 months from baseline.
  Sleep-wake patterns were evaluated using actigraphy. The children were asked to wear an actigraphy watch (MotionWatch 8, CamNtech, UK), which monitors movement and light exposure, for 5-7 days. Fragmentation Index (index units) is used to measure sleep quality, composed of the percentage of measured mobile time and immobile bouts with a duration ≤1 min, during assumed sleep.
Actigraphy to evaluate sleep-wake patterns: Wake Bouts (seconds) | Will be conducted at baseline (time of enrollment) and again 1-3 months after completion of the physical exercise intervention, within 6 months from baseline.
  Sleep-wake patterns were evaluated using actigraphy. The children were asked to wear an actigraphy watch (MotionWatch 8, CamNtech, UK), which monitors movement and light exposure, for 5-7 days. Wake bouts (seconds) means single episodes of wakefulness during the sleep period. Total daytime activity score (score units) was defined by the sum of the activity counts during wakefulness..
Actigraphy to evaluate sleep-wake patterns: Total Activity Score (score units) | Will be conducted at baseline (time of enrollment) and again 1-3 months after completion of the physical exercise intervention, within 6 months from baseline.
  Actigraphy to evaluate sleep-wake patterns: Wake Bouts (seconds) Description: Sleep-wake patterns were evaluated using actigraphy. The children were asked to wear an actigraphy watch (MotionWatch 8, CamNtech, UK), which monitors movement and light exposure, for 5-7 days. Total daytime activity score (score units) was defined by the sum of the activity counts during wakefulness.
Autism Spectrum Screening Questionnaire (ASSQ) | Will be conducted at baseline (time of enrollment) and again 1-3 months after completion of the physical exercise intervention, within 6 months from baseline.
  ASSQ is a screening questionnaire for autism spectrum disorder, containing 27 questions or statements assessing behaviors related to ASD. The ratings available are "no" (0 point), "somewhat" (1 point), "yes" (2 points). The points are added up to a total score of maximum 54 points. For a clinical population the score 19 are used as a cutoff to indicate autism spectrum disorder.
Behavior Rating Inventory of Executive Function , Second Edition (BRIEF-2) | Will be conducted at baseline (time of enrollment) and again 1-3 months after completion of the physical exercise intervention, within 6 months from baseline.
  BRIEF measuring executive functions and self-regulation in children and adolescents ages 5-18 in the parent form. The questionnaire consists of 63 statements and nine clinical scales: inhibition, self-monitor, shift, emotional control, initiate, working memory, plan/organize, task-monitor and organizing of materials. These scales are distributed under three domains: behavioral index, emotional index and cognitive index. The global executive composite (GEC) averages all assessment values. The rater records their answer via a Likert-type format N (never), S (sometimes) or O (often). Results are presented in T-score format (M=50, SD=10) and a higher T-score suggests that the child exhibits significant difficulties with executive functions. The results could also be compared to age-matched norms. Cut-off scores: 60-64 mildly elevated; 65-69 potentially clinically elevated; ≥70 clinically elevated difficulties.
Child Sensory Profile (CSP) | Will be conducted at baseline (time of enrollment) and again 1-3 months after completion of the physical exercise intervention, within 6 months from baseline.
  CSP is an assessment to evaluate a child's sensory processing patterns in different environments and how they impact on daily functioning. The parent form can be used for children ages 3-14 years. It consists of 86 statements and the parent record their answer by choosing between "almost always", "frequently", "half of the time", "occasionally", "almost never" or "does not apply". Most of the items are counted under one of the quadrants: seeking (the degree to which a child obtains sensory input), avoiding (the degree to which a child is bothered by sensory input), sensitivity (the degree to which a child detects sensory input) and registration (the degree on which a child misses sensory input). The form also provides information about how the child processes different modalities of sensory inputs divided into the following sensory sections: auditory, visual, touch, movement, body position and oral. Behavioral responses related to sensory inputs are divided into the following behavior
Social Responsiveness Scale (SRS) | Will be conducted at baseline (time of enrollment) and again 1-3 months after completion of the physical exercise intervention, within 6 months from baseline.
  SRS aims to identify social impairment associated with ASD and quantify its severity. The school age form applies for parents to children and adolescents ages 4-18 years. It consists of 65 items which are rated on a graduated response scale: "never true", "sometimes true", "often true" and "almost always true". Five subscales are used for evaluating treatment: social awareness, social cognition, social communication, social motivation and restricted interest and repetitive behavior. The subscales are preferably not used for screening or diagnosis. The total and subscale scores are compared to clinical cut-offs indicating presence of autism-related social impairments; 60-75 mild to moderate social impairment; ≥76 severe social impairment.
Strengths and Difficulties Questionnaire (SDQ) | Will be conducted at baseline (time of enrollment) and again 1-3 months after completion of the physical exercise intervention, within 6 months from baseline
  SDQ is an emotional and behavioral screening questionnaire for parents to children and adolescents ages 4-17 years. It consists of 33 questions or statements and the responder records their answer for the first 25 items on the response scale: "not true", "somewhat true" or "certainly true". The remaining items address the severity and the duration of the difficulties. The first 25 items asses five scales: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems and prosocial behavior. The total score helps to categorize the child or adolescent as having "normal", "borderline" or "abnormal" difficulties. For the subscales there are clinical cut-off scores.
Swanson, Nolan, and Pelham 26-item Rating Scale (SNAP-IV) | Will be conducted at baseline (time of enrollment) and again 1-3 months after completion of the physical exercise intervention, within 6 months from baseline.
  SNAP-IV is a 30-item rating scale for parents to assess symptoms of ADHD (inattention and hyperactivity/impulsivity) and symptoms of oppositional defiant disorder, based on the DSM criteria. It is divided into subscales for inattention, hyperactivity/impulsivity, and oppositional behavior. Symptom severity is rated on a 4-point scale: not at all (0), just a little (1), quite a bit (2) and very much (3). Subscale scores are calculated and compared to clinical cut-off scores. ≥ 1.67 indicates clinical difficulties for combinated inattention + hyperactivity/impulsivity.
Cognitive testing with CANTAB: Intra-Extra Dimensional Set Shift (IED) | Will be conducted at baseline (time of enrollment) and again 1-3 months after completion of the physical exercise intervention, within 6 months from baseline.
  For cognitive assessment, all children underwent a selection of tests from the computerized Cambridge Neuropsychological Test Automated Battery (CANTAB). IED includes 27 outcome measures to evaluate rule acquisition and reversal, requiring visual discrimination, attentional set formation, maintenance, shifting, and attention flexibility. The participant must work out a rule that determines which stimulus is correct. After six correct responses, the stimuli and/or rule changes. Outcome measure assess the number of stages completed, the numbers of trials completed, the number of errors made and response latency.
  Outcome measurements as they are described in CANTAB Connect Research: Admin Application User Guide, Cambridge Cognition limited 2022, V1.25. Note that each test has several more outcome measurements that we excluded in our analysis.
Cognitive testing with CANTAB: Paired Association Learning (PAL) | Will be conducted at baseline (time of enrollment) and again 1-3 months after completion of the physical exercise intervention, within 6 months from baseline.
  For cognitive assessment, all children underwent a selection of tests from the computerized Cambridge Neuropsychological Test Automated Battery (CANTAB). With 21 outcome measures, the PAL test evaluates visual memory and new learning abilities. Boxes are displayed and one or more of them contains a pattern. The patterns are then displayed in the middle and the participant must select the box containing the same pattern. Outcome measurements are stages completed, memory scores, the errors made, and the number of trials required to locate the patterns.
Cognitive testing with CANTAB: Reaction Time (RTI) | Will be conducted at baseline (time of enrollment) and again 1-3 months after completion of the physical exercise intervention, within 6 months from baseline.
  Comprising 21 outcome measures, this test assesses motor and mental response speed, as well as movement time, reaction time, response accuracy, and impulsivity. The participant must select and hold a button while circles are presented on the screen. When a circle with a yellow dot in it appears, the participant must react as fast as possible and select the circle with the dot in it. Outcome measures are reaction time and movement time.
Cognitive testing with CANTAB: Stockings of Cambridge (SOC) | Will be conducted at baseline (time of enrollment) and again 1-3 months after completion of the physical exercise intervention, within 6 months from baseline.
  Featuring 27 outcome measures, the SOC test assesses spatial planning and problem-solving strategy formulation. The participant is requested to move balls to copy a pattern and use as few moves as possible. Movement time is discounted in a part of the task where the participants just copy the movements made by the computer which mimics the movements the participant made when solving the original problem. Outcome measures include difficulty level reached, mean moves used and thinking time.
Cognitive testing with CANTAB: Spatial Working Memory (SWM) | Will be conducted at baseline (time of enrollment) and again 1-3 months after completion of the physical exercise intervention, within 6 months from baseline.
  The SWM test, with 24 outcome measures, assesses the retention and manipulation of visuospatial information, providing measures of strategy use and working memory. The participant is requested to select the boxes and using a process of elimination to find a token in each of a number of boxes. The number of boxes gradually increases, and the color and position of the boxes changes between trials. Outcome measures include different type of errors and strategy.
Evaluation of the intervention | After completion of the intervention, within 6 months from baseline.
  Semi-structured or structured interviews with participants and/or parents.
Sleep Electroencephalogram (EEG): Posterior Dominant Rhythm (Hz) | Will be conducted at baseline (time of enrollment) and again 1-3 months after completion of the physical exercise intervention, within 6 months from baseline.
  Participants will undergo a sleep EEG recording lasting approximately 40 minutes to assess brain electrical activity during sleep, to measure posterior Dominant Rhythm in Hertz (Hz), which is the main background alpha frequency.
Sleep Electroencephalogram (EEG): Interictal epileptiform activity (IEA) | Will be conducted at baseline (time of enrollment) and again 1-3 months after completion of the physical exercise intervention, within 6 months from baseline.
  Participants will undergo a sleep EEG recording lasting approximately 40 minutes to assess brain electrical activity during sleep, to measure IEA; the frequency of interictal epileptiform activity was assessed and graded as rare, moderate, or frequent.
Sleep Electroencephalogram (EEG): Sleep Spindles (counts) | Will be conducted at baseline (time of enrollment) and again 1-3 months after completion of the physical exercise intervention, within 6 months from baseline.
  Participants will undergo a sleep EEG recording lasting approximately 40 minutes to assess brain electrical activity during sleep, to measure sleep spindles; number of sleep spindles during the first 5 minutes following the first vertex wave, as well as after the occurrence of the first sleep spindle after sleep onset.

CONTACTS AND LOCATIONS:
Overall Officials: Christine T Ekdahl, Associate professor, Principal Investigator — Div. Clinical Neurophysiology, Dept Clinical Sciences, Lund University & Clinical Neurophysiology, Department of Medical Imaging and Physiology, Skåne University Hospital, Lund, Sweden.
Locations (1):
- Div. Clinical Neurophysiology, Dept Clinical Sciences, Lund University, SE-221 85 Lund, Sweden, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data. This is an exploratory study with a small number of participants, and sharing the data could potentially compromise participant confidentiality.